CLINICAL TRIAL: NCT02603276
Title: Lipid-lowering Effect of Phytosterols, Red Yeast Rice and Their Combination in Moderately Hypercholesterolemic Subjects in Primary Prevention for Cardiovascular Diseases: a Randomized, Double Blind, Clinical Trial
Brief Title: Lipid-lowering Effect of Phytosterols, Red Yeast Rice and Their Combination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Full professor of internal medicine, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PhytoRed
Record Dates: First submitted 2015-08-27; First posted 2015-11-11 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; dietary supplements; red yeast rice; plant sterols
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols; red yeast rice

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Plant sterols (Active Comparator): Plant sterols 800 mg per dose, 1 liquid stick per day, per 8 weeks
  Interventions: Dietary Supplement: Plant sterols
- Red Yeast Rice (Active Comparator): Red Yeast Rice 200 mg containing 5 mg monacolin K per daily dose, 1 liquid stick per day, per 8 weeks
  Interventions: Dietary Supplement: Red Yeast Rice
- Red Yeast Rice plus Plant sterols (Experimental): lant sterols 800 mg per dose + Red Yeast Rice 200 mg containing 5 mg monacolin K per daily dose, 1 liquid stick per day, per 8 weeks
  Interventions: Dietary Supplement: Plant sterols; Dietary Supplement: Red Yeast Rice plus Plant sterols

INTERVENTIONS:
Dietary Supplement: Plant sterols — Plant sterols 800 mg/dose, 1 liquid stick per day, for 8 weeks
  Arms: Plant sterols; Red Yeast Rice plus Plant sterols
Dietary Supplement: Red Yeast Rice — Red Yeast Rice titrated in 5 mg monacolin K per daily dose, 1 liquid stick per day, for 8 weeks
  Arms: Red Yeast Rice
Dietary Supplement: Red Yeast Rice plus Plant sterols — Red Yeast Rice titrated in 5 mg monacolin K per daily dose plus Plant sterols 800 mg/dose, together in 1 liquid stick per day, for 8 weeks
  Arms: Red Yeast Rice plus Plant sterols

SUMMARY:
A large body of evidence confirm the cholesterol lowering effect of phytosterols and red yeast rice. Because their mechanisms of action mime the ones of chemical statins and cholesterol absorption inhibitors, it is plausible that their association will provide a more relevant (and safe) LDL cholesterolemia reduction.

DETAILED DESCRIPTION:
A large body of literature suggest that the patients are strongly interested in self-medicating them with "natural" products aimed at reducing their plasma level of LDL-cholesterol. Plant sterols and red yeast rice are among the most widely marketed product with these properties in Western countries. However plant sterols per se have a limited effect on cholesterolemia, while full dosed red yeast rice can induce myalgias and myopathies as statins do. In this context, the aim of the investigators' study was to evaluate if the association of both products at low dosage could induce an additive or synergistic effect in term of LDL-reduction in humans.

ELIGIBILITY:
Inclusion Criteria:

* LDL-cholesterolemia between 130 and 190 mg/dL

Exclusion Criteria:

* Type 2 diabetes
* Previous cardiovascular disease
* Assumption of lipid-lowering drugs or dietary supplements
* Previous intolerance to red yeast rice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
LDL cholesterolemia reduction from baseline and between groups | 8 weeks
  Absolute and % reduction of LDL cholesterolemia after 8 weeks of treatment

SECONDARY OUTCOMES:
Non-HDL cholesterolemia reduction from baseline and between groups | 8 weeks
  Absolute and % reduction of of non-HDL cholesterolemia after 8 weeks of treatment
Number of Participants With Treatment-Related Adverse Events | 8 weeks
  Subjective tolerability of the tested treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Principal Investigator — University of Bologna
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Italy

REFERENCES:
- [Result] Cicero AFG, Fogacci F, Rosticci M, Parini A, Giovannini M, Veronesi M, D'Addato S, Borghi C. Effect of a short-term dietary supplementation with phytosterols, red yeast rice or both on lipid pattern in moderately hypercholesterolemic subjects: a three-arm, double-blind, randomized clinical trial. Nutr Metab (Lond). 2017 Sep 25;14:61. doi: 10.1186/s12986-017-0214-2. eCollection 2017. PMID 29021813